CLINICAL TRIAL: NCT02191709
Title: A Phase I, Single Dose, Controlled Two-way Crossover Study to Evaluate the Relative Bioavailability of Orally Administered Dextromethorphan Syrup (21 mg Dextromethorphan Hydrobromide Monohydrate) in Comparison to Dextromethorphan Soft Pastilles (21 mg Dextromethorphan Hydrobromide Monohydrate) in Healthy Male and Female Subjects Who Are Extensive Metabolisers for Cytochrom P450 (CYP) 2D6
Brief Title: Relative Bioavailability of Dextromethorphan Syrup in Comparison to Dextromethorphan Soft Pastilles in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1134.2
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- Dextromethorphan syrup (Experimental): Bisoltussin® Syrup
  Interventions: Drug: Dextromethorphan syrup
- Dextromethorphan soft pastilles (Active Comparator): Silomat® DMP soft pastilles
  Interventions: Drug: Dextromethorphan soft pastilles

INTERVENTIONS:
Drug: Dextromethorphan syrup
  Arms: Dextromethorphan syrup
Drug: Dextromethorphan soft pastilles
  Arms: Dextromethorphan soft pastilles

SUMMARY:
Study to investigate the relative bioavailability of orally administered dextromethorphan syrup in comparison to dextromethorphan (DMP) soft pastilles in healthy male and female subjects who are extensive metabolisers for CYP 2D6

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), clinical laboratory tests
* Age ≥18 and Age ≤55 years
* BMI ≥18.5 and BMI ≤30 kg/m2 (Body Mass Index)
* Extensive metabolisers for CYP 2D6
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or which prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within one month prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for TdP (Torsades de points) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

For female subjects:

* Pregnancy or planning to become pregnant within 2 months of study completion
* Positive pregnancy test
* No adequate contraception in women of childbearing potential during the study, i.e. sterilization, intrauterine device, hormonal contraception
* Lactation period

Exclusion criteria specific for this study:

* Use of drugs that inhibit or induce cytochrome P 450 enzymes, especially CYP 2D6, within 30 days prior to first administration of the study medication or during the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-01; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) - for dextromethorphan and dextrorphan (total and free) | predose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 32 hours after drug administration
Cmax (maximum measured concentration of the analyte in plasma) - for dextromethorphan and dextrorphan (total and free) | predose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 32 hours after drug administration
tmax (time from dosing to the maximum measured concentration of the analyte in plasma) - for dextromethorphan and dextrorphan (total and free) | predose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 32 hours after drug administration

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) - all analytes | predose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 32 hours after drug administration
AUCt1-t2 (Area under the concentration time curve of the analyte in plasma over the time interval t1 to t2) - all analytes | predose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 32 hours after drug administration
%AUCtz-∞ (percentage of the AUC0-∞ that is obtained by extrapolation) - all analytes | predose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 32 hours after drug administration
λz (terminal rate constant in plasma) - all analytes | predose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 32 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) - all analytes | predose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 32 hours after drug administration
MRTpo (mean residence time of the analyte in the body after oral administration) - all analytes | predose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 32 hours after drug administration
CL/F (apparent clearance of the analyte in the plasma after oral administration) - all analytes | predose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 32 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an oral dose) - all analytes | predose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 32 hours after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) - 3-hydroxy-morphinan (total and free) and 3- methoxy-morphinan | predose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 32 hours after drug administration
Cmax (maximum measured concentration of the analyte in plasma) - 3-hydroxy-morphinan (total and free) and 3- methoxy-morphinan | predose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 32 hours after drug administration
tmax (time from dosing to the maximum measured concentration of the analyte in plasma) - 3-hydroxy-morphinan (total and free) and 3- methoxy-morphinan | predose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 32 hours after drug administration
Number of patients with adverse events | up to 53 days
Number of patients with abnormal changes in laboratory parameters | Screening, 14 days after the end of last treatment period
Number of patients with abnormal changes in 12-lead ECG (electrocardiogram) (including QT interval and heart rate corrected QTcF and QTcB) | Screening, Day 1, 14 days after the end of last treatment period
Number of patients with clinically significant changes in vital signs (blood pressure (BP), pulse rate (PR)) | Screening, Day 1, 14 days after the end of last treatment period
Assessment of tolerability on a 4-point scale | Day 2 of each treatment period